CLINICAL TRIAL: NCT05966935
Title: Effect of Fenugreek and Cumin Powder on Anthropometric Indices of Overweight and Obese Adults
Brief Title: Effect of Fenugreek and Cumin Powder on Overweight and Obese People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Veterinary and Animal Sciences, Lahore - Pakistan (Other)
Responsible Party: Principal Investigator, Sanaullah Iqbal, Professor, University of Veterinary and Animal Sciences, Lahore - Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fenugreek and cumin powder
Record Dates: First submitted 2023-07-14; First posted 2023-08-01 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Overweight and Obesity
Keywords: Fenugreek powder; Cumin powder; Body Composition; Anthropometric Indices
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Participants will be divided into two groups. One group will receive the Fenugreek Cumin Powder. The other group will not receive the powder
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fenugreek cumin powder (Experimental): Overweight and Obese adults in this group will receive fenugreek cumin powder daily twice a day before morning and evening meals for 8 weeks
  Interventions: Combination Product: Fenugreek Cumin Powder
- Control group (No Intervention): Overweight and obese participants in this group will not receive fenugreek and cumin powder or any intervention for 8 weeks

INTERVENTIONS:
Combination Product: Fenugreek Cumin Powder — Fenugreek and Cumin seeds will be procured from the market. They will be cleaned of debris, winnowed, and grinded to fine powder passed through a mesh size of 30 for metal cleaning. 5g of fenugreek powder and 5g of cumin powder will be packed in packets. Participants in the intervention group will be instructed to consume the powder before breakfast and dinner with a glass of water.
  Arms: fenugreek cumin powder

SUMMARY:
The objective of this study is to investigate the effect of fenugreek and cumin powder on the anthropometric indices of overweight and obese adults aged 18-30 years. This study design intends to answer following question:

Will fenugreek and cumin powder mixture result in change of anthropometric measurements {Body Mass Index[BMI], Waist-Hip Ratio, Fat Mass

DETAILED DESCRIPTION:
Obesity is a chronic disorder of carbohydrate and lipid metabolism and is characterized by an increased fat deposition in adipose tissue and other internal organs .

Obesity leads to the development of insulin resistance, type-2 diabetes, coronary heart disease, cancer, respiratory disease, and osteoarthritis. The World Obesity Atlas 2022 predicts that one billion people globally, including 1 in 5 women and 1 in 7 men, will be living with obesity by 2030.

Pakistan ranks tenth out of 188 countries, with 50% of population overweight or obese Several studies have investigated the effect of fenugreek and cumin supplementation on anthropometric measures but the findings have been inconsistent. Only few studies directly focused on powder supplementation. The study aims to investigate the effect of fenugreek and cumin powder supplementation on body measurements for weight loss. This will help in developing a rather inexpensive, herbal mixture for weight loss.

Galactomannan present in fenugreek capture and excrete sugars from body before it moves in the blood, this causes the loss of weight The percent gain in body weight was significantly low in groups supplemented with fenugreek Cumin improves anthropometric indices in overweight. Cumin powder reduced weight, Body Mass Index[BMI], waist circumference, fat mass and percentage significantly.

This study consists of following phases Phase 1: Fenugreek and cumin powder preparation Phase 2: 30 Participants will be recruited after filling the consent form and screened through a questionnaire throughout the university. Individuals with Body Mass Index[BMI] >23kg/m2, Waist-Hip-Ratio >0.8 will be recruited in the study after fulfilling the criterion (patients of thyroid, Polycystic ovary syndrome[PCOS], Hypertension[HTN] will be excluded). Participants not following any fitness regime or specific diet will be recruited further. Baseline body measurements will be taken by inbody analyzer. They will be given powder packed in packets to be used for 8 weeks twice a day before breakfast and dinner. Experimental Design : Overweight and obese adults will be assigned to two groups ( Intervention group and control). Participants will be requested to record the following information daily: Consumption of FCP( fenugreek cumin powder) and any side effects if experienced after consumption.

The control group will not receive powder or any other intervention. Phase 3: Measurements will be taken after intervention

Statistical Analysis:

Microsoft excel will be used for data coding. Descriptive analysis will be done by using SPSS[Statistical Package for Social Sciences] version 23( SPSS for windows version 23; SPSS Inc., Chicago).

Independent sample t-test and Pearson chi-square will be performed to compare the treatment and control groups. P value < 0.05 will be considered significant for all analysis.

ELIGIBILITY:
Inclusion Criteria:

* overweight and obese( BMI>23 kg/m^2)

Exclusion Criteria:

* pregnant women
* Thyroid
* PCOS
* HTN
* fitness regime
* specific diet

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-12-28 (Actual)

PRIMARY OUTCOMES:
weight change in kilograms | change from baseline weight after 2 months
  Electronic weighing scale will be used to assess weight change in both groups
Change in Body fat mass in kilograms and percentages | change from baseline readings after 2 months
  body fat mass and percentage will be assessed through inbody analyzer 270
Change in BMI in kg/m^2 | change from baseline reading after 2 months
  the BMI will be calculated using weight(kg) and height(m^2)
Change in Waist- Hip Ratio | change from baseline reading after 2 months
  the WHR will be calculated using inbody analyzer 270

SECONDARY OUTCOMES:
Change in Basal metabolic Rate( BMR) | Change from baseline after 2 months
  The BMR will be calculated using Inbody analyzer 270
change in Protein mass of body (grams) | change from baseline reading after 2 months
  this protein mass will be assessed through Inbody analyzer 270

CONTACTS AND LOCATIONS:
Overall Officials: Sanaullah Iqbal, PhD, Principal Investigator — University of Veterinary and Animal Sciences Lahore, Punjab
Locations (1):
- University of Veterinary and Animal Sciences, Lahore, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khosla P, Gupta DD, Nagpal RK. Effect of Trigonella foenum graecum (Fenugreek) on blood glucose in normal and diabetic rats. Indian J Physiol Pharmacol. 1995 Apr;39(2):173-4. PMID 7649611
- [Background] Geberemeskel GA, Debebe YG, Nguse NA. Antidiabetic Effect of Fenugreek Seed Powder Solution (Trigonella foenum-graecum L.) on Hyperlipidemia in Diabetic Patients. J Diabetes Res. 2019 Sep 5;2019:8507453. doi: 10.1155/2019/8507453. eCollection 2019. PMID 31583253
- [Background] Hameed S, Arshad MS, Ahmad RS, Hussain G, Imran M, Arshad MU, Ahmed A, Imran M, Imran A. Potential preventive and protective perspectives of different spice powders and their mixtures in rat model. Lipids Health Dis. 2020 Apr 23;19(1):78. doi: 10.1186/s12944-020-01223-9. PMID 32326942
- [Background] Khateeb S, Albalawi A, Alkhedaide A. Regulatory effect of diosgenin on lipogenic genes expression in high-fat diet-induced obesity in mice. Saudi J Biol Sci. 2021 Jan;28(1):1026-1032. doi: 10.1016/j.sjbs.2020.11.045. Epub 2020 Nov 18. PMID 33424396
- [Background] Kumar P, Bhandari U, Jamadagni S. Fenugreek seed extract inhibit fat accumulation and ameliorates dyslipidemia in high fat diet-induced obese rats. Biomed Res Int. 2014;2014:606021. doi: 10.1155/2014/606021. Epub 2014 Apr 29. PMID 24868532
- [Background] Laudadio V, Nasiri-Dehbaneh M, Bilal RM, Qotbi A, Javandel F, Ebrahimi A, Seidavi A, Slozhenkina M, Gorlov I, Dunne PG, Tufarelli V. Effects of different levels of dietary black cumin (Nigella sativa L.) and fenugreek (Trigonella foenum-graecum L.) and their combination on productive traits, selected blood constituents, microbiota and immunity of broilers. Anim Biotechnol. 2022 Oct;33(5):941-954. doi: 10.1080/10495398.2020.1853138. Epub 2020 Dec 16. PMID 33325302
- [Background] Mathern JR, Raatz SK, Thomas W, Slavin JL. Effect of fenugreek fiber on satiety, blood glucose and insulin response and energy intake in obese subjects. Phytother Res. 2009 Nov;23(11):1543-8. doi: 10.1002/ptr.2795. PMID 19353539
- [Background] Tavakoli-Rouzbehani OM, Faghfouri AH, Anbari M, Nikpayam O, PourMirzaei Olyaei H, Alizadeh M. Efficacy of Cuminum Cyminum supplementation on lipid profile and anthropometric parameters: A systematic review and meta-analysis of randomized controlled clinical trials. Phytother Res. 2022 Jan;36(1):380-394. doi: 10.1002/ptr.7327. Epub 2021 Nov 25. PMID 34825421
- [Background] Peng Y, Sun Q, Xu W, He Y, Jin W, Yuan L, Gao R. Vitexin ameliorates high fat diet-induced obesity in male C57BL/6J mice via the AMPKalpha-mediated pathway. Food Funct. 2019 Apr 1;10(4):1940-1947. doi: 10.1039/c9fo00148d. Epub 2019 Mar 15. PMID 30874277
- [Background] Said O, Saad B, Fulder S, Khalil K, Kassis E. Weight loss in animals and humans treated with "weighlevel", a combination of four medicinal plants used in traditional arabic and islamic medicine. Evid Based Complement Alternat Med. 2011;2011:874538. doi: 10.1093/ecam/nen067. Epub 2011 Jun 16. PMID 18952688
- [Background] Sharma MS, Choudhary PR. Effect of Fenugreek Seeds Powder (Trigonella foenum-graecum L.) on Experimental Induced Hyperlipidemia in Rabbits. J Diet Suppl. 2017 Jan 2;14(1):1-8. doi: 10.3109/19390211.2016.1168905. Epub 2016 Apr 12. PMID 27070043
- [Background] Yadav UC, Baquer NZ. Pharmacological effects of Trigonella foenum-graecum L. in health and disease. Pharm Biol. 2014 Feb;52(2):243-54. doi: 10.3109/13880209.2013.826247. Epub 2013 Oct 9. PMID 24102093